CLINICAL TRIAL: NCT00592969
Title: Evaluation of Efficacy and Safety of Metformin Plus Biphasic Insulin Aspart or Insulin NPH in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Metformin Plus Biphasic Insulin Aspart 30 in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1570
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Metformin; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: metformin
Drug: biphasic insulin aspart

SUMMARY:
This trial is conducted in South America. The aim of this trial is to evaluate the efficacy of metformin plus biphasic insulin aspart or insulin NPH on blood glucose control in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with insulin NPH or are insulin-naive
* Body mass index (BMI) below 35.0 kg/m2
* HbA1c between 7.5-11.0%

Exclusion Criteria:

* Participation in any other clinical trial involving investigational products within the last 3 months
* History of drug or alcohol dependence
* Known impaired hepatic function
* Known or suspected allergy to human insulin NPH, insulin aspart or any component of the composition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2003-12-03 (Actual); Primary Completion 2004-11-02 (Actual); Study Completion 2004-11-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 12 weeks of treatment

SECONDARY OUTCOMES:
PPBG values
Glucose profiles
Hypoglycemia
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Mariano Acosta S/n, Argentina
- Novo Nordisk Investigational Site, Santa Efigênia, Brazil

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com